CLINICAL TRIAL: NCT06565182
Title: The Acute Effect of Physical Exercise in Pregnancy on the Fetoplacental Unit: A Randomized Crossover Trial Comparing Aerobic Versus Resistance Exercise
Brief Title: The Acute Effect of Physical Exercise in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EDGE002233
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Related
Keywords: blood flow; pregnancy; aerobic exercise; resistance exercise; doppler ultrasound; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous aerobic exercise (Experimental): The continuous aerobic intervention was performed on a bicycle in a seated position at a moderate exercise intensity. Heart rate and RPE was implemented to ensure moderate intensity level. The participants were allowed to warm up for 5 minutes before starting to cycle at the predetermined HR ranges for 25 minutes. The total duration of exercise was 30 minutes.
  Interventions: Other: Exercise
- Resistance exercise (Experimental): The acute resistance intervention consisted of four exercises performed using Technogym equipment at a moderate intensity. Every exercise consisted of 3 sets of 20 repetitions, with 1 minute rest in between sets, equaling 30 minutes of exercise in total. The four exercises were performed using the following Technogym devices: vertical traction, chest press, low row, leg press. Prior to the start of each exercise, a short maximal resistance test provided by the Technogym equipment was executed to determine moderate intensity.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The intervention consists of two different types of moderate intensity exercise: Continuous aerobic and resistance exercise.

SUMMARY:
The goal of this crossover clinical trial is to investigate the acute physiological effect of exercise on the uterine and fetal blood flow in pregnancy. The main questions it aims to answer are:

* What is the acute physiological effect of exercise on the uterine and fetal blood flow in pregnancy?
* What is the acute physiological effect of continuous aerobic exercise versus resistance exercise on the uterine and fetal blood flow in pregnancy?
* What is the effect of physical activity levels on the uterine and fetal blood flow in pregnancy?

Researchers will compare the continuous aerobic exercise to the resistance exercise with a 3-6-week interval to examine the acute physiological effect on the uterine and fetal blood flow.

Participants will:

* Fill in a physical activity level questionnaire at baseline.
* Complete either continuous aerobic exercise or resistance exercise and take blood flow measurements.
* Complete the remaining type of exercise after a 3-6-week interval and take blood flow measurements.

ELIGIBILITY:
Inclusion Criteria:

* pregnant, over the age of 18 years, singleton pregnancy, both primigravidas and multigravidas, uncomplicated pregnancy and absence of contra-indications for exercise as per Canadian guidelines (Mottola et al. 2018).

Exclusion Criteria:

* smoking, substance abuse, chronic diseases, fetal growth restriction, fetal abnormalities, hypertension, history of premature delivery, vaginal hemorrhage, placenta previa, contractions before/during intervention, diabetes mellitus, preeclampsia and previous pregnancy complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Blood flow using doppler ultrasound measurements | The measurements were taken before and after each exercise bout. Participants rested for at least 15 minutes before their baseline measurement was evaluated. Reassessment was done within 15 minutes after the intervention.
  Measurements of the pulsatility index of the left and right uterine artery, umbilical artery and middle cerebral artery were taken using Doppler ultrasound. The pulsatility indexes were determined by taking the average of three waveforms from the Doppler velocity measurements.

SECONDARY OUTCOMES:
Physical activity levels | Physical activity levels were assessed at baseline.
  Physical fitness levels were assessed using the Dutch version of the IPAQ-SF questionnaire. Categorical scores are defined as low, moderate and high physical activity levels. The category labeled 'high' is classified when vigorous-intensity activity on at least 3 days achieves a minimum of at least 1500 MET-minutes/week or 7 or more days of any combination of walking, moderate-intensity or vigorous-intensity activities achieve a minimum of at least 3000 MET-minutes/week on total physical activity. 'Moderate' is classified if vigorous-intensity activity is performed for at least 20 minutes per day on 3 or more days; or moderate-intensity activity and/or walking is performed at least 30 minutes per day for 5 or more days; or 5 or more days of any combination of walking, moderate intensity or vigorous-intensity activities achieve a total physical activity of at least 600 MET minutes/week. All who do not meet the criteria for 'moderate' or 'high' are assigned to the category 'low'.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No